CLINICAL TRIAL: NCT04485091
Title: Association of Trichloroacetic Acid Peel With Photobiomodulation in the Treatment of Skin Photoaging of the Hands: a Study Protocol for a Controlled, Randomized, Double-blind Clinical Trial.
Brief Title: TCA Peel and Photobiomodulation for Hand Rejuvenation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Co-supervisor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHOTOACID
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Skin Aging
Keywords: Photoaging; Photodamage; Chemical peel; Photobiomodulation; Phototherapy; Skin rejuvenation; Rejuvenation of hands; low-level laser therapy (LLLT); light emitting diode (LED)
MeSH Terms: interventions — phytobacteriomycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: 20% TCM and PBM (Experimental): 21 participants will be included in this group. Application of chemical peel of 20% trichloroacetic acid solution (TCM) in association with photobiomodulation (PBM) with red spectrum LED (660nm) on the back of the hands.
  Interventions: Combination Product: 20% TCM and PBM
- Group B: 20% TCM and PBM placebo (Placebo Comparator): 21 participants will be included in this group. Application of chemical peel of 20% trichloroacetic acid solution (TCM) in association with simulated photobiomodulation on the back of the hands.
  Interventions: Other: 20% TCM and PBM placebo

INTERVENTIONS:
Combination Product: 20% TCM and PBM — The chemical peel (20% TCM) will be carried out monthly, totaling 04 sessions. The application of photobiomodulation (PBM) will start shortly after the observation of frosting level I, which characterizes an exfoliation of superficial depth. Although the application sessions take place monthly, medical evaluations will be carried out fortnightly for the other orientations, filling in scales and photographs. For the PBM, a LED device with an irradiance of 10 milliwatts per square centimeter (mW/cm²) in continuous operation mode and a wavelength of 660 nm will be used. It will provide an energy density of 4 J/cm² within 400 seconds of irradiation.
  Arms: Group A: 20% TCM and PBM
Other: 20% TCM and PBM placebo — The chemical peel (20% TCM) will be carried out monthly, totaling 04 sessions. The application of photobiomodulation (PBM) will be simulated soon after the observation of frosting level I. The patient will not be aware of the simulation of the procedure. Although the application sessions take place monthly, medical evaluations will be carried out fortnightly for the other orientations, filling in scales and photographs.
  Arms: Group B: 20% TCM and PBM placebo

SUMMARY:
Photodamage is a growing concern in contemporary society because promotes early skin aging and different pathologies resulting from prolonged and repeated exposure to ultraviolet solar radiation, which is considered the main extrinsic factor of this process. Affected by radiation, the hands play an important role in the manifestation and visibility of aging, as they are very exposed body regions. The study proposal is developed by the potential mechanism of tissue repair, skin rejuvenation, anti-inflammatory and analgesic effects of photobiomodulation, complementing the benefits of chemical peel. The main objective of this randomized, controlled, double-blind clinical trial is to compare the photorejuvenating effects of 20% trichloroacetic acid (TCM) peel applied alone and the effects of the association of 20% TCM peel with 660nm light emitting diode (LED) photobiomodulation (PBM) in the treatment of the back of the hands. Participants will be divided into 2 groups and will receive different therapies according to the allocation group. Group A will be subjected to 04 chemical peel sessions of 20% TCM and PBM. Group B will also receive the 04 chemical peel sessions of 20% TCM with PBM simulation. The application sessions will be monthly and the consultations for fortnightly evaluations. Analysis of photoaging characteristics such as fine and coarse wrinkles, dyschromias and global assessment of the back of the hands will be carried out using periodic standardized photographs. A visual-analog pain scale and a 5-point Likert scale will also be applied regularly to assess participants' satisfaction.

DETAILED DESCRIPTION:
Participants will be divided into two groups for the treatment of photoaging of hands:

(A) Group 20% TCM + PBM: Application of chemical peel of 20% trichloroacetic acid solution in association with photobiomodulation with red spectrum LED (660nm) on the back of the hands.

(B) Group 20% TCM + PBM placebo: Application of chemical peel of 20% trichloroacetic acid solution in association with simulated photobiomodulation on the back of the hands.

It is observed that all participants included in the study will receive treatment recommended for photoaging on the back of the hands. The chemical peel (20% TCM solution) will be performed monthly, totaling 04 sessions with an average time of 40 minutes (guidelines, photos, skin exfoliation) with intervals of 04 weeks between applications. Biweekly assessments (guidelines and photos) will be carried out with an average time of 20 minutes during the study period. In addition, a group will also be subjected to photobiomodulation with 660nm LED during the sessions for the analysis of the association of therapies and comparison with exfoliation monotherapy.

It is noteworthy that both hands will be treated and control will be maintained in another randomized and uniform group, with no possibility of ethical compromise of different therapies with asymmetric results in the participants. Another important benefit provided by the separation of the control group will be the impossibility of light to influence the non-irradiated tissue. This case would occur if the hand subjected to photobiomodulation plus exfoliation was in the same individual as the hand subjected to exfoliation monotherapy. This influence is defended by countless scientists who research on the systemic effects of phototherapy.

In addition, both groups will prepare the skin properly before the treatments in order to enhance the effects of the exfoliation, allow the uniform penetration of the chemical solution in the back of the hands, decrease the healing time after the procedure and significantly reduce the risks of major complications such as post-inflammatory hyperpigmentation. Throughout the period, the participants will also be instructed on the importance of photoprotection with the daily use of factor 30 sunscreen. If there is a patient with severe hypersensitivity or major complications, the intervention will be discontinued immediately and properly treated according to its severity.

It should be noted that regardless of the results obtained at the end of the research, even if photobiomodulation improves or accelerates the benefits of chemical peeling, participants will not be submitted to new treatment sessions, as both groups will already receive treatment recommended for photoaging of hands. Furthermore, the application of photobiomodulation without the association of previous skin exfoliation is unlikely to bring better results, because early application after tissue injury is the most important factor for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Individuals without comorbidities or with controlled comorbidities (ASA I and ASA II physical status classification).
* Participants must also have skin phototype I, II or III according to the Fitzpatrick classification.

Exclusion Criteria:

* Smoking, alcoholic, oncological, malnourished, anemic, pregnant, immunosuppressed participants.
* Patients with blood dyscrasias, psychiatric illnesses, collagen diseases (even with proper control), photosensitivity, individuals undergoing chemotherapy or hormone therapy and with scar changes (keloids and hypertrophic scar).
* Also excluded from the study are individuals who performed previous aesthetic procedures on their hands and use of medications that influence skin color, such as amiodarone, tetracyclines, tricyclic antidepressants, phenothiazines and others.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Fine wrinkles | 6 months
  The back of both hands of the participants will be photographed before starting the skin preparation for the experiments (day 0). Standardized photo sessions according to the Clinical Photography Committee of the Plastic Surgery Educational Foundation will also take place in each biweekly medical evaluation to monitor the evolution of photorejuvenation. All photographs will be evaluated after 30 days of the last treatment session by 02 independent experts in 04 distinct clinical signs about photoaging: fine wrinkles, coarse wrinkles, abnormal pigmentation and global evaluation. The global evaluation is used to have a general impression of the photodamage, as shown by Mckenzie, 2011. The 04 clinical signs will be characterized separately by a scale from 0 to 9, with 0 representing the absence of changes and 9 representing the maximum of changes. The Kappa coefficient will be used to measure agreement between the examiners.

SECONDARY OUTCOMES:
Coarse wrinkles | 6 months
  The back of both hands of the participants will be photographed before starting the skin preparation for the experiments (day 0). Standardized photo sessions according to the Clinical Photography Committee of the Plastic Surgery Educational Foundation will also take place in each biweekly medical evaluation to monitor the evolution of photorejuvenation. All photographs will be evaluated after 30 days of the last treatment session by 02 independent experts in 04 distinct clinical signs about photoaging: fine wrinkles, coarse wrinkles, abnormal pigmentation and global evaluation. The global evaluation is used to have a general impression of the photodamage, as shown by Mckenzie, 2011. The 04 clinical signs will be characterized separately by a scale from 0 to 9, with 0 representing the absence of changes and 9 representing the maximum of changes. The Kappa coefficient will be used to measure agreement between the examiners.
Abnormal pigmentation | 6 months
  The back of both hands of the participants will be photographed before starting the skin preparation for the experiments (day 0). Standardized photo sessions according to the Clinical Photography Committee of the Plastic Surgery Educational Foundation will also take place in each biweekly medical evaluation to monitor the evolution of photorejuvenation. All photographs will be evaluated after 30 days of the last treatment session by 02 independent experts in 04 distinct clinical signs about photoaging: fine wrinkles, coarse wrinkles, abnormal pigmentation and global evaluation. The global evaluation is used to have a general impression of the photodamage, as shown by Mckenzie, 2011. The 04 clinical signs will be characterized separately by a scale from 0 to 9, with 0 representing the absence of changes and 9 representing the maximum of changes. The Kappa coefficient will be used to measure agreement between the examiners.
Global evaluation | 6 months
  The back of both hands of the participants will be photographed before starting the skin preparation for the experiments (day 0). Standardized photo sessions according to the Clinical Photography Committee of the Plastic Surgery Educational Foundation will also take place in each biweekly medical evaluation to monitor the evolution of photorejuvenation. All photographs will be evaluated after 30 days of the last treatment session by 02 independent experts in 04 distinct clinical signs about photoaging: fine wrinkles, coarse wrinkles, abnormal pigmentation and global evaluation. The global evaluation is used to have a general impression of the photodamage, as shown by Mckenzie, 2011. The 04 clinical signs will be characterized separately by a scale from 0 to 9, with 0 representing the absence of changes and 9 representing the maximum of changes. The Kappa coefficient will be used to measure agreement between the examiners.
Visual Analog Scale (VAS) for pain | 6 months
  The visual analog scale has been used to measure intangible quantities such as pain, quality of life and anxiety, since the 1920s. Measuring the subjective experience of pain is a continuous challenge in medicine, and VAS, despite its limitations, is a primary outcome measure validated for pain intensity. Participants will use the scale to measure pain intensity during the study during biweekly medical evaluations. The number 0 means the total absence of pain complaints, while the number 10 is equivalent to the greatest pain ever experienced by the participant.
Scale of Satisfaction | 6 months
  Monthly, participants will be evaluated at the specialty clinic to analyze the results provided by the study. The individuals will answer a questionnaire composed by a 5-point Likert scale modified by the author about the satisfaction of the obtained results

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Momolli, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho (UNINOVE), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishida-Yamamoto A, Kartasova T, Matsuo S, Kuroki T, Iizuka H. Involucrin and SPRR are synthesized sequentially in differentiating cultured epidermal cells. J Invest Dermatol. 1997 Jan;108(1):12-6. doi: 10.1111/1523-1747.ep12285611. PMID 8980279
- [Background] Zhang S, Duan E. Fighting against Skin Aging: The Way from Bench to Bedside. Cell Transplant. 2018 May;27(5):729-738. doi: 10.1177/0963689717725755. Epub 2018 Apr 25. PMID 29692196
- [Background] Blanpain C, Fuchs E. Epidermal stem cells of the skin. Annu Rev Cell Dev Biol. 2006;22:339-73. doi: 10.1146/annurev.cellbio.22.010305.104357. PMID 16824012
- [Background] Soleymani T, Lanoue J, Rahman Z. A Practical Approach to Chemical Peels: A Review of Fundamentals and Step-by-step Algorithmic Protocol for Treatment. J Clin Aesthet Dermatol. 2018 Aug;11(8):21-28. Epub 2018 Aug 1. PMID 30214663
- [Background] Lindley LE, Stojadinovic O, Pastar I, Tomic-Canic M. Biology and Biomarkers for Wound Healing. Plast Reconstr Surg. 2016 Sep;138(3 Suppl):18S-28S. doi: 10.1097/PRS.0000000000002682. PMID 27556760
- [Background] Yaar M, Gilchrest BA. Photoageing: mechanism, prevention and therapy. Br J Dermatol. 2007 Nov;157(5):874-87. doi: 10.1111/j.1365-2133.2007.08108.x. Epub 2007 Aug 17. PMID 17711532
- [Background] Avci P, Gupta A, Sadasivam M, Vecchio D, Pam Z, Pam N, Hamblin MR. Low-level laser (light) therapy (LLLT) in skin: stimulating, healing, restoring. Semin Cutan Med Surg. 2013 Mar;32(1):41-52. PMID 24049929
- [Result] McKenzie NE, Saboda K, Duckett LD, Goldman R, Hu C, Curiel-Lewandrowski CN. Development of a photographic scale for consistency and guidance in dermatologic assessment of forearm sun damage. Arch Dermatol. 2011 Jan;147(1):31-6. doi: 10.1001/archdermatol.2010.392. PMID 21242389